CLINICAL TRIAL: NCT06296862
Title: Effect of Dietary Approaches to Stop Hypertension Diet on Heart Failure Status in Older Adults
Brief Title: Effect of DASH on HF Outcomes Heart Failure Status in Older Adults (DASH HF)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Collaborators: Emory University (Other)
Responsible Party: Principal Investigator, Elisabeth Lilian Pia Sattler, Ph.D., B.S. Pharm, Assistant Professor, University of Georgia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005563
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Dietary Approaches To Stop Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary Approaches to Stop Hypertension Diet (Experimental)
  Interventions: Other: Dietary Approaches to Stop Hypertension Diet
- Usual Diet (No Intervention)

INTERVENTIONS:
Other: Dietary Approaches to Stop Hypertension Diet — The DASH diet is a heart-healthy eating pattern that is focused on adequate consumption of fruits, vegetables, whole grains, low-fat dairy, fish, poultry, beans, nuts, and vegetables oils while emphasizing limited intake of foods containing saturated fat, such as fatty red meats, full-fat dairy products, and tropical oils, such as coconut, palm kernel, and palm oils, as well as sugar-sweetened beverages and sweets. The chosen 4 week intervention duration phase is consistent with previous research showing positive effects of consuming a sodium-reduced dietary intervention on volume status and is longer than in other studies showing positive effects of DASH diet consumption on cardiac outcomes among HF patients. Potential carryover effects are minimized by a washout period of 4 weeks. The meal plan has been previously developed based on NHLBI guidelines for the DASH diet.
  Arms: Dietary Approaches to Stop Hypertension Diet

SUMMARY:
The purpose of this study is to examine the effect of the Dietary Approaches to Stop Hypertension (DASH) diet has on heart failure status in older adults. This study is important because it may provide a low-cost strategy to help reduce hospitalizations and deaths for heart failure patients. Participants will be adults age 65 and older with heart failure. They will have 4 study visits, each lasting about 2 hours, and will be in the study for 12 weeks. They will also be asked about their dietary consumption 6 times, each time lasting about 45 minutes. All in-person study visits will take place in the Emory GCRC. Participants will have physical exams, body measurements, blood tests, urinalysis, chart review, and answer surveys. They will be randomized to eat only the DASH diet provided to them for 4 weeks either at the beginning or end of their participation in the study. Participants will be recruited from heart failure patients at Emory University Hospital, Emory University Hospital Midtown, and Emory Outpatient Advanced Heart Failure Therapy Center. The total enrollment planned under Emory's oversight, accounting for screen failures and withdrawals, will be n=38 participants. The study team will obtain informed consent prior to the first study visit either in person, or, alternatively, over the phone, if requested by participants. Specimens and data obtained in this study will not be banked for future use.

ELIGIBILITY:
Inclusion Criteria:

* 65+ years of age
* Heart failure diagnosis and symptoms, as outlined by the 2021 European Society of Cardiology diagnostic guidelines
* Residence within 50 miles of Emory University
* Have undergone hemodynamic monitoring device implantation (CardioMEMS, Abbott)
* Have received optimized HF therapy for 3+ months post CardioMEMS implantation

Exclusion Criteria:

* Heart failure-related hospitalization or heart failure medication changes within 1 month
* Renal disease stages IV-V
* Expected survival < 12 months
* Dementia or Alzheimer's disease
* Limited English literacy and communication skills

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
B-natriuretic peptide (BNP) | Study visit 1-4
  Clinically relevant natriuretic peptide

SECONDARY OUTCOMES:
N-terminal-proBNP (NT-proBNP) | Study visit 1-4
  Clinically relevant natriuretic peptide
Systolic and Diastolic Pulmonary Artery Pressures | Patient-driven measurement data points during intervention/control phase (8 weeks)
  Early indicator of heart failure complications

CONTACTS AND LOCATIONS:
Locations (1):
- Emory Clinical Cardiovascular Research Center (ECCRI), Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No